CLINICAL TRIAL: NCT00543205
Title: A Pharmacokinetic Study of Genasense® (Bcl-2 Antisense Oligonucleotide) in Combination With Dacarbazine (DTIC) in Subjects With Advanced Melanoma and Normal or Impaired Hepatic Function
Brief Title: Pharmacokinetics of G3139 in Subjects With Advanced Melanoma, Including Those With Normal Hepatic Function and Those With Moderate Hepatic Impairment
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated due to very slow enrollment
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPK103
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2009-03

CONDITIONS: Advanced Melanoma and Normal or Impaired; Hepatic Function
MeSH Terms: interventions — oblimersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Genasense® (G3139, oblimersen sodium) — Genasense 7 mg/kg/day for 5 days
  Other Names: G3139; Oblimersen; Oblimersen sodium

SUMMARY:
This is an open-label, parallel-group study with a total of 16 evaluable subjects. Subjects will be assigned to 1 of the following cohorts: Cohorts I (subjects with normal hepatic function; n+8 and Cohort II (subjects with moderate hepatic impairment, Child-Pugh classification Grade B; n=8). If, for any reason, the Genasense infusion is interrupted or discontinued prior to completion or the rate of administration of the Genasense infusion is changed, the subject will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant melanoma
* Metastatic Stage IV disease, or Stage III disease that is not surgically resectable
* ECOG Performance status of 0,1,or 2
* Adequate venous access
* Agreement to practice effective methods of birth control
* Hepatically impaired consistent with Child-Pugh classification Grade B

Exclusion Criteria:

* Chronic intravascular coagulopathy confirmed by the presence of fibrinogen degradation products, metastases to the liver, or exudative ascites
* Prior organ allograft
* Requirement for concomitant anticoagulant therapy (with the exception of 1 mg/day of warfarin for central line prophylaxis) while receiving protocol therapy
* Known hypersensitive to DTIC
* Prior treatment with Genasense

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of G3139 | 6-day period

SECONDARY OUTCOMES:
Safety | 30 days post last dose of study medication